CLINICAL TRIAL: NCT00669058
Title: Study for Dermatological Evaluation of Topic Compatibility (Primary and Accumulated Dermical Irritability, Dermical Sensitivity) of Dermacyd Tina Gel Tangerina Mix.
Brief Title: Dermatological Evaluation of Topic Compatibility-Dermacyd Tina Gel Tangerina Mix
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: GMA-CO/Medical Director, sanofi-aventis administrative office France
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LACAC_L_03736
Record Dates: First submitted 2008-04-23; First posted 2008-04-29 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Healthy
Keywords: hygiene
MeSH Terms: interventions — Lactic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Lactic acid (Dermacid)

SUMMARY:
The purpose of this study is to demonstrate the absence of irritation potential (primary dermic irritability and cumulated dermic irritability) and allergy (sensibilization) of the product Dermacyd Tina Gel Tangerina Mix

ELIGIBILITY:
Inclusion Criteria:

* Phototype Skin I,II, III e IV
* Integral skin test in the region

Exclusion Criteria:

* Lactation or gestation
* Use of Antiinflammatory and/or immunosuppression drugs
* Personnel history of atopy
* History of sensitivity or irritation for topic products
* Active cutaneous disease
* Use of new drugs or cosmetics during the study

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2007-12; Primary Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
The absence of primary and accumulated dermal irritability and dermal sensitivity will be evaluated using International Contact Dermatitis Research Group (ICDRG) scale. | six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, Study Director — Sanofi-aventis administrative office Brazil
Locations (1):
- Sanofi-aventis administrative office, São Paulo, São Paulo, Brazil